CLINICAL TRIAL: NCT05553145
Title: The Prevalence of Autoimmune Antibodies in Patients with Type 2 Diabetes Managed by Endocrinology Vs. Primary Care
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-797
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients Seen by their Endocrinologist: Patients whose diabetes is managed by their Endocrinologist
  Interventions: Diagnostic Test: Autoimmune Antibody Assays
- Patients Seen by their Primary Care Provider: Patients whose diabetes is managed by their Primary Care Provider
  Interventions: Diagnostic Test: Autoimmune Antibody Assays

INTERVENTIONS:
Diagnostic Test: Autoimmune Antibody Assays — GAD-65, Islet cell-Ab, IA-2 Ab, anti-insulin Ab, and ZnTn8 Ab

SUMMARY:
The purpose of this study is to assess the levels of autoimmune markers of diabetes in those with a type 2 diabetes diagnosis.

DETAILED DESCRIPTION:
Autoimmune markers can appear when the body uses its natural defense system to mistakenly attack the patient's own cells because it cannot tell the difference between the patient and foreign cells. The study investigators want to determine if there are any differences in these marker levels when comparing patients who are managed by their primary care provider and patients managed by endocrinology. Patients will be asked to come in for a blood draw. This sample will be used for autoimmune antibody testing. An antibody is a protein in the blood that is made to find and respond to a specific antigen. An antigen is something that triggers the body to have an immune response. Patient participation in the research study will last for the duration of one visit to the clinic for informed consent and a blood draw.

The clinical implications of detecting this type of diabetes can be profound, as it can identify patients who are at risk of becoming insulin dependent in the near future, and therefore may require a change in diabetes management to avoid adverse outcomes. In addition, identifying these patients may also open up the door for treatments directed at stopping the complete autoimmune destruction of insulin producing cells, potentially delaying or avoiding the need for insulin dependency.

The study team presumes that autoimmune markers of diabetes will be detected in patients with a diagnosis of type 2 diabetes and the prevalence of these markers will be higher among patients managed by endocrinology. The population of patients found to have detectable autoimmune markers of diabetes will differ from the population of patients without these markers. The population of patients managed by endocrinology that are found to have detectable autoimmune markers of diabetes will differ from the population of patients managed by primary care. The population of patients with more than 1 autoimmune antibody are more likely to require insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Language: English
* Age: ≥ 18
* Type 2 diabetes
* Ability to provide informed consent before any trial-related activities. Trial-related activities are any procedure that would not have been performed during normal management of the subject.

Exclusion Criteria:

* Patients with a diagnosis of T1D or LADA in their problem list
* Patients with an encounter diagnosis for T1D or LADA
* Mental incapacity or language barrier (non-English speaking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from community hospital either coming in to see their primary care physician or endocrinologist.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of autoimmune antibodies in patients with Type 2 Diabetes | One-time blood draw at consent/screening
  Percentage of subjects with T2D and detectable autoimmune antibodies calculated as the percentage of subjects that test positive for at least one of the autoimmune antibodies

SECONDARY OUTCOMES:
Prevalence of autoimmune antibodies in patients with T2D managed by endocrinology | One-time blood draw at consent/screening
  Percentage of subjects whose diabetes is managed by an endocrinologist with T2D and detectable autoimmune antibodies calculated as the percentage of subjects that test positive for at least one of the autoimmune antibodies
Prevalence of autoimmune antibodies in patients with T2D managed by primary care | One-time blood draw at consent/screening
  Percentage of subjects whose diabetes is managed by a primacy care physician with T2D and detectable autoimmune antibodies calculated as the percentage of subjects that test positive for at least one of the autoimmune antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pantalone, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Twinsburg Family Health & Surgery Center, Twinsburg, Ohio, United States